CLINICAL TRIAL: NCT06959875
Title: Different Methods in Therapeutic Communication Training for Student Nurses in the Perinatal Loss: High-Fidelity Simulation and Paper - Pencil Simulation
Brief Title: Therapeutic Communication Training in Perinatal Loss: Simulation-Based Approaches
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Acibadem University (Other)
Responsible Party: Principal Investigator, Merve Coskun, Assistant professor, Acibadem University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2025/05-188
Record Dates: First submitted 2025-04-16; First posted 2025-05-07 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-04

CONDITIONS: Simulation-based Learning; Communication Skills; Paper-Pencil Simulation; High-fidelity Simulation

STUDY DESIGN:
Intervention Model Description: Parallel Assignment Randomized Controlled Experimental Design
Who Masked: Participant
Masking Description: In the single-blind method, subjects do not know which of the experimental or control groups they were selected and therefore which method was applied to them. The researcher knows the subjects selected for the experimental and control groups, and therefore which method was applied to which subjects.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-Fidelity Simulation-Based Therapeutic Communication Training (Experimental): Participants in this group engaged in a high-fidelity simulation scenario involving perinatal loss, using a realistic clinical setting with mannequins and role-play. The simulation aimed to provide an experiential learning environment that fosters emotional engagement and realistic practice of therapeutic communication techniques. Students received a structured debriefing session following the simulation.
  Interventions: Behavioral: High-Fidelity Simulation-Based Therapeutic Communication Training
- Paper-Pencil Simulation-Based Therapeutic Communication Training (Active Comparator): Participants in this group participated in a paper-pencil simulation that presented a written clinical scenario involving perinatal loss. Students were asked to analyze the situation, write down appropriate therapeutic communication responses, and discuss these in a guided session. This method focused on the cognitive application of theoretical knowledge in a reflective and structured manner.
  Interventions: Behavioral: Paper-Pencil Simulation-Based Therapeutic Communication Training

INTERVENTIONS:
Behavioral: High-Fidelity Simulation-Based Therapeutic Communication Training — This intervention involves a structured, high-fidelity simulation scenario in a clinical skills lab setting using mannequins and standardized patients. The scenario focuses on communication with a patient experiencing perinatal loss. The session includes pre-briefing, simulation, and debriefing components.
  Arms: High-Fidelity Simulation-Based Therapeutic Communication Training
Behavioral: Paper-Pencil Simulation-Based Therapeutic Communication Training — This intervention utilizes a written clinical case scenario related to perinatal loss. Students read the scenario and write appropriate therapeutic communication responses, followed by group discussion and instructor feedback. The focus is on reflection and theoretical integration.
  Arms: Paper-Pencil Simulation-Based Therapeutic Communication Training

SUMMARY:
This study aims to evaluate the effect of simulation-based education on nursing students' therapeutic communication skills in managing perinatal loss. Perinatal loss, defined as early fetal loss before 20 weeks of gestation and late fetal loss at or after 20 weeks, is a traumatic experience that significantly impacts parents, especially mothers, on biological, psychological, social, and spiritual levels. Prolonged grief reactions can lead to complicated grief, anxiety, depression, hopelessness, and relationship disturbances. Nursing students are trained to adopt a biopsychosocial approach in patient care and are expected to support grieving individuals by normalizing emotions, identifying coping strategies, and facilitating healthy grief processing. Simulation is recognized as an effective teaching method in developing communication and therapeutic skills among nursing students. This research investigates how simulation-based training can enhance students' therapeutic communication competencies when supporting individuals experiencing perinatal loss.

ELIGIBILITY:
Inclusion Criteria:

* Completion of the theoretical course on postpartum care in the Women's Health and Diseases Nursing course.
* Successful completion of the Human Behavior and Communication course.
* Completion of training on perinatal grief and therapeutic communication skills prior to the simulation training.

Exclusion Criteria:

* Medical or Psychological Conditions Impacting Communication
* Incomplete Training or Lack of Pre-Simulation Education
* Inability to Participate in the Debriefing Session
* Language Barriers

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-01-30 (Actual); Study Completion 2025-01-30 (Actual)

PRIMARY OUTCOMES:
Therapeutic Communication Skills Performance | Immediately during scenario completion (Day 1)
  Students' ability to effectively demonstrate therapeutic communication skills during a simulated patient encounter involving perinatal loss. Assessed using the Therapeutic Communication with Patients Experiencing Perinatal Loss Simulation Application Checklist, which evaluates competencies such as providing presence, empathy, active listening, calming guidance, providing psychological support, and applying therapeutic communication techniques. Performance is rated as "Yes," "Partially," or "No" based on observed behaviors.
Perceived Communication Skills Self-Assessment | Immediately before debriefing session (Day 1)
  Students' self-evaluation of their communication abilities following the simulation experience, measured by the Communication Skills Assessment Form. This form covers 20 communication techniques, both therapeutic and nontherapeutic, rated on a 10-point scale, with higher scores reflecting stronger perceived communication competencies.
Student Satisfaction and Self-Confidence in Learning Scale (SCLS) | Immediately after debriefing session (Day 1)
  Students' level of satisfaction with the simulation-based learning experience and their self-confidence in applying learned skills, assessed through the Student Satisfaction and Self-Confidence in Learning Scale (SCLS). The scale includes two subdimensions-Student Satisfaction and Self-Confidence in Learning-measured via a 5-point Likert scale. Higher scores indicate greater satisfaction with the simulation and higher confidence in using therapeutic communication skills.
Simulation Execution Checklist Evaluation | During scenario execution (Day 1)
  The degree to which the simulation was implemented according to planned steps and standards. This outcome measures the fidelity, completeness, and quality of the simulation process itself, as evaluated by observers using a checklist. It ensures consistency, scenario realism, and adherence to key components critical for achieving the intended learning objectives.

SECONDARY OUTCOMES:
Reflection on Learning and Communication Effectiveness | Immediately after debriefing session (Day 1)
  Students' ability to critically reflect on their learning experiences and assess the effectiveness of their communication during the simulation. Reflection focuses on recognizing strengths and areas for improvement in therapeutic communication, understanding emotional responses during patient interactions, and identifying strategies for enhancing future clinical practice. This outcome promotes self-awareness, deeper learning, and the internalization of communication skills through structured debriefing and written or verbal reflections.

CONTACTS AND LOCATIONS:
Locations (1):
- Merve Coşkun, Ataşehir, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will be stored in an online database (e.g., Mendeley). Data will be available upon request after the study results are published by the researchers.

REFERENCES:
- [Background] Adib-Rad H, Basirat Z, Faramarzi M, Mostafazadeh A, Bijani A. Psychological distress in women with recurrent spontaneous abortion: A case-control study. Turk J Obstet Gynecol. 2019 Sep;16(3):151-157. doi: 10.4274/tjod.galenos.2019.88899. Epub 2019 Oct 10. PMID 31673466
- [Background] Graneheim UH, Lundman B. Qualitative content analysis in nursing research: concepts, procedures and measures to achieve trustworthiness. Nurse Educ Today. 2004 Feb;24(2):105-12. doi: 10.1016/j.nedt.2003.10.001. PMID 14769454
- [Background] Hanshaw SL, Dickerson SS. High fidelity simulation evaluation studies in nursing education: A review of the literature. Nurse Educ Pract. 2020 Jul;46:102818. doi: 10.1016/j.nepr.2020.102818. Epub 2020 Jun 9. PMID 32623148
- [Background] Herbert D, Young K, Pietrusinska M, MacBeth A. The mental health impact of perinatal loss: A systematic review and meta-analysis. J Affect Disord. 2022 Jan 15;297:118-129. doi: 10.1016/j.jad.2021.10.026. Epub 2021 Oct 20. PMID 34678403
- [Background] Kang SJ, Kim Y. The Impact of Perinatal Loss Nursing Simulation among Undergraduate Students. Int J Environ Res Public Health. 2022 Jul 14;19(14):8569. doi: 10.3390/ijerph19148569. PMID 35886421
- [Background] Kim J, Park JH, Shin S. Effectiveness of simulation-based nursing education depending on fidelity: a meta-analysis. BMC Med Educ. 2016 May 23;16:152. doi: 10.1186/s12909-016-0672-7. PMID 27215280
- [Background] Leyland A, Choucri L. Student midwives' lived experiences of caring for bereaved parents following perinatal loss using actor-based simulation: A phenomenological study. Midwifery. 2024 Mar;130:103913. doi: 10.1016/j.midw.2023.103913. Epub 2024 Jan 10. PMID 38241799
- [Background] Li YY, Au ML, Tong LK, Ng WI, Wang SC. High-fidelity simulation in undergraduate nursing education: A meta-analysis. Nurse Educ Today. 2022 Apr;111:105291. doi: 10.1016/j.nedt.2022.105291. Epub 2022 Feb 3. PMID 35158134
- [Background] Rudland JR, Golding C, Wilkinson TJ. The stress paradox: how stress can be good for learning. Med Educ. 2020 Jan;54(1):40-45. doi: 10.1111/medu.13830. Epub 2019 Sep 11. PMID 31509282